CLINICAL TRIAL: NCT05185752
Title: Comparative Analysis of Three Locoregional Anesthesia Methods in Breast Tumour Pathology Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ref. 070/2018
Record Dates: First submitted 2021-11-16; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2020-05

CONDITIONS: Postoperative Pain; Chronic Post Operative Pain; Breast Tumor; Locoregional Anesthesia; Breast Pain
Keywords: ESP block; PECS block; SIFP block; breast tumor surgery; locoregional anesthesia
MeSH Terms: conditions — Pain, Postoperative; Breast Neoplasms; Mastodynia

STUDY DESIGN:
Intervention Model Description: Patients undergoing breast tumour surgery were randomised to undergo one of three locoregional techniques in three study groups (Erector Spinae Plane block -ESP block-, Pectoral Nerve Block type II -PECS II block-, or Serratus-Intercostal fascial Plane Block-SIFP block). Locoregional techniques were performed under light sedation and then, general anaesthesia was used for the breast tumour surgery.
Who Masked: Participant
Masking Description: The type of masking applied was:
  First part of study (until 24 hours after surgery): single-blind, the patient did not know what type of treatment he had received, but the anaesthesiologist in the operating room, and the main intraoperative and immediate postoperative period evaluator were aware of all this.
  Second part of study (3 months and 1 year after surgery): double-blind, the patient did not know what type os treatment he had received, and the anesthesiologist who was the responsible of collecting data through the telephone interview or her medical history, did not know the treatment taken by the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Erector Spinae Plane Block (ESP block) (Active Comparator): The patient is positioned in the prone position, the probe is used to locate in cross-section the T4 spinous process. Next, using a lateral scan, approximately 3 cm away, the costotransverse joint is located, and then change to sagittal ultrasound vision. By locating the intertransverse line with the probe, the following anatomical structures can be identified: three longitudinal muscles (trapezius, rhomboid, erector spinae).
  The needle enters in a single punction at an angle of 45º, in the cranio-caudal direction, until it touches the apex of the costotransverse image. Subsequently, 30 cc of 0.25% bupivacaine are administered in the depth of the erector spinae, which will remain elevated.
  Interventions: Procedure: ESP block: Locoregional Interfascial Anesthesic Technique
- Pectoral Nerve type II Block (PECS II block) (Active Comparator): The patient is positioned supine, with the ipsilateral upper limb extended. The clavicular external third line is drawn. In parallel, the lower costal line and the infraclavicular space are highlighted. The probe obtains an image that allows the identification of the pectoralis major and pectoralis minor.
  If colour Doppler is added, the acromiothoracic artery is identified and must be avoided.
  The needle enters at an angle of 45º from medial to lateral, and 20 cc of 0.25% bupivacaine are administered. Next, needle advances in the interfascial space between the pectoral minor and serratus anterior and 10 cc of 0.25% bupivacaine are administered.
  Interventions: Procedure: PECS II block: Locoregional Interfascial Anesthesic Technique
- Serratus-Intercostal Fascial Plane Block (SIFP block) (Active Comparator): The patient is positioned supine, with the ipsilateral upper extremity at a 90º angle. The fourth, fifth, and sixth intercostal spaces are identified in the mid-axillary line. In coronal section, it is possible to appreciate the subcutaneous cellular tissue, the serratus anterior, and the intercostal muscles.
  The needle is introduced at an angle of 30º. From caudal to cranial and resting the needle on the fourth rib, 30 cc of 0.25% bupivacaine are administered between the serratus anterior and lateral intercostal muscles.
  Interventions: Procedure: SIFP Block Locoregional Interfascial Anesthesic Technique

INTERVENTIONS:
Procedure: SIFP Block Locoregional Interfascial Anesthesic Technique — Interfascial blocks emerged as locoregional techniques that incorporate ultrasonography to visualise the anatomy while administrating the drug, reducing the rate of complications. There are multiple locoregional interfascial techniques continue to be implemented; in 2011 Blanco described Pectoral Nerve Block (PECS block); in 2012, Serratus-Intercostal Fascial Plane Block (SIFP) was described, and in 2016, Forero described the Erector Spinae Plane Block (ESP).
  Drug: 30 cc 0.25% bupivacaine. Nerves blocked by SIFP block: lateral and anterior cutaneous branches of the 2nd-6th Intercostal Nerves.
  Devices: S-Nerve® ultrasound was used in all three techniques; linear 6 to 13 Megahertz and convex 2 to 5 Megahertz transducers and 22G (Gauge) x 50 mm needles.
  Arms: Serratus-Intercostal Fascial Plane Block (SIFP block)
Procedure: PECS II block: Locoregional Interfascial Anesthesic Technique — Interfascial blocks emerged as locoregional techniques that incorporate ultrasonography to visualise the anatomy while administrating the drug, reducing the rate of complications. There are multiple locoregional interfascial techniques continue to be implemented; in 2011 Blanco described Pectoral Nerve Block (PECS block); in 2012, Serratus-Intercostal Fascial Plane Block (SIFP) was described, and in 2016, Forero described the Erector Spinae Plane Block (ESP).
  Drug: 30 cc 0.25% bupivacaine. Nerves blocked by PECS-II: Lateral Pectoral Nerve and Medial Pectoral Nerve Devices: S-Nerve® ultrasound was used in all three techniques; linear 6 to 13 Megahertz and convex 2 to 5 Megahertz transducers and 22G (Gauge) x 50 mm needles.
  Arms: Pectoral Nerve type II Block (PECS II block)
Procedure: ESP block: Locoregional Interfascial Anesthesic Technique — Interfascial blocks emerged as locoregional techniques that incorporate ultrasonography to visualise the anatomy while administrating the drug, reducing the rate of complications. There are multiple locoregional interfascial techniques continue to be implemented; in 2011 Blanco described Pectoral Nerve Block (PECS block); in 2012, Serratus-Intercostal Fascial Plane Block (SIFP) was described, and in 2016, Forero described the Erector Spinae Plane Block (ESP).
  Drug: 30 cc 0.25% bupivacaine. Nerves blocked by ESP Block: dorsal and ventral branch block of the spinal nerves; white and gray communicating branches of the sympathetic nerves that go to the thoracic sympathetic chain.
  Devices: S-Nerve® ultrasound was used in all three techniques; linear 6 to 13 Megahertz and convex 2 to 5 Megahertz transducers and 22G (Gauge) x 50 mm needles.
  Arms: Erector Spinae Plane Block (ESP block)

SUMMARY:
The present study compares the Erector Spinae Plane (ESP) block, Pectoral (PECS II) block, and Serratus-Intercostal Fascial Plane (SIFP) block. This is the first article to compare these three locoregional nerve block techniques in acute and chronic postoperative pain in breast tumour surgery.

From June 1, 2018, to June 30, 2019, 103 patients undergoing breast cancer surgery were randomised to undergo one of three locoregional techniques (35 for ESP block, 34 for PECS II block, 34 for SIFP block). Locoregional techniques were performed under light sedation and then, general anaesthesia was used for the breast cancer surgery. Outcomes measured included pain (visual analog scale [VAS] in immediate postoperatory and at 24 hours. It also was collected opioid use at 24 hours, adverse events, and length of stay (for acute postoperatory). Moreover, at 3 months, a telephone interview was conducted with the patient and VAS was questioned. A year later, the patient was questioned again and asked for VAS, location of her pain, and pharmacological treatment. It was collected if patients were assisted or not by a Pain Unit.

DETAILED DESCRIPTION:
Introduction

Breast surgery, armpit surgery, and the possible addition of reconstructive surgery lead to acute postoperative pain. Anaesthesiology aims to manage this pain adequately, with locoregional anaesthesia as a key tool in constant evolution.

In 2011, Blanco described the Pectoral Nerve Block (PECS). Interfascial blocks emerged as locoregional techniques that incorporate ultrasonography to visualise the anatomy while administrating the drug, reducing the rate of complications. Since then, multiple locoregional interfascial techniques continue to be implemented; in 2012, Serratus-Intercostal Fascial Plane Block (SIFP) was described, and in 2016, Forero described the Erector Spinae Plane Block (ESP).

However, there is little literature that compares the various blocks that exist. The investigators conducted a literature search in PubMed, Cochrane, and clinicaltrials.gov, with a study period from January 2011 to February 2021. The descriptors used were Erector Spinae Plane Block AND Breast, Pectoral Block AND Breast, Intercostal Nerve Block AND Breast, Locoregional Anaesthesia AND Breast, Serratus Anterior Plane Block AND Breast Surgery. The inclusion criteria were: studies with female patients, related to surgical intervention of breast tumour pathology, including every type of surgery, and publications in English or Spanish. The exclusion criteria were: studies of another type of locoregional anaesthesia; studies that do not separately evaluate the efficacy of the block but add more than one locoregional anaesthetic technique; studies with purely anatomical purposes (in cadaver, radiological, experimental animal model); and research on pharmacological issues. A total of 917 references were obtained, and after applying the different filters, this was reduced to 11 publications. These studies conclude that acute postoperative pain management is better when supplementing the patient with locoregional technique than without locoregional anaesthesia.

Moreover, chronic postoperative pain (CPP) in breast tumour surgery has an overall incidence of 25-30% one year after the intervention. The best established risk factor for CPP is having suffered severe and uncontrolled postoperative acute pain (PAP) as well as the existence of preoperative pain, requiring large consumption of analgesia in the perioperative period. Actually, 10-50% of postoperative patients with pain will develop CPP. An adequate approach of PAP reduces the risk of CPP.

There is literature enough to affirm that supplementing patients with locoregional technique to general anesthesia for breast tumour surgery, gets a better pain control than only undergoing general anesthesia. However, there is a lack of literature comparing the effectiveness of applying interfascial locoregional techniques, and it is unknown which one of them could be more recommended to prevent CPP.

Approval by the Ethics Committee

This controlled clinical trial was approved by the Ethics Committee for Research with Medicines of the Institut d'Investigació Sanitària Pere Virgili (IISPV) in Tarragona, Spain (Ref. 070/2018 dated May 31, 2018). The principles of the Helsinki Declaration were respected. Written informed consent was obtained from every patient.

Sample Size

The sample size was determined in the study design by the IISPV so that it was appropriate for the objectives set and assuming the particular conditions. The calculation was performed with a public software called GRANMO, version 7.12, for analysis of variances after reviewing the literature. Accepting an alpha risk of 0.05 and beta risk of less than 0.2 in bilateral contrast, 34 subjects were necessary for each of the three groups to detect a minimum difference of 2 points on the Visual Analogue Scale (VAS) and a standard deviation of 2.4. A loss to follow-up rate of 10% was considered.

Period of study

During the 13-month period (from June 1, 2018 to June 30, 2019), 165 patients underwent breast cancer surgery, of which 103 were included in the present study.

Population assigned to the health department corresponding to the Verge de la Cinta Hospital in Tortosa (Tarragona) that underwent elective surgery for breast tumor pathology.

Methodology

Hypothesis

The initial hypothesis of the study proposes that the Erector Spinae Plane Block (ESP) confers better control of acute postoperative pain and less chronic postoperative pain than the other two more common locoregional anesthesia methods (Pectoral Nerve Block type II -PECS II block- or Serratus-Intercostal Fascial Plane block -SIFP block).

Masking and Randomization

Randomisation was carried out by blocks in a 1: 1: 1 ratio, avoiding numerical inequality between the treatment groups. In this way, the patient was incorporated into block 1 (ESP), next patient to block 2 (PECS II), and the next patient to block 3 (SIFP).

The type of masking applied was:

First part of study (until 24 hours after surgery): single-blind, the patient did not know what type of treatment he had received, but the anaesthesiologist in the operating room, and the main intraoperative and immediate postoperative period evaluator were aware of all this.

Second part of study (3 months and 1 year after surgery): double-blind, the patient did not know what type os treatment he had received, and the anesthesiologist who was the responsible of collecting data through the telephone interview or her medical history, did not know the treatment taken by the patient.

The variables taken into account were:

Age Body mass index Tumour size Visual Analogue Scale (VAS) score Pathological diagnosis Tumour staging Type of surgery.

Anesthetic Procedure

All patients were monitored with pulse oximetry (SpO2), a six-lead electrocardiogram, and non-invasive blood pressure. The corresponding locoregional technique was performed under light sedation with IV midazolam 0.015-0.03 mg / kg and supplemental oxygen with nasal cannulas. S-Nerve® ultrasound was used in all three techniques; linear 6 to 13 Megahertz and convex 2 to 5 Megahertz transducers and 22G (Gauge) x 50 mm needles.

Erector Spinae Plane block (ESP block):

The patient is positioned in the prone position, the probe is used to locate in cross-section the T4 spinous process. Next, using a lateral scan, approximately 3 cm away, the costotransverse joint is located, and then change to sagittal ultrasound vision. By locating the intertransverse line with the probe, the following anatomical structures can be identified: three longitudinal muscles (trapezius, rhomboid, erector spinae).

The needle enters in a single punction at an angle of 45º, in the cranio-caudal direction, until it touches the apex of the costotransverse image. Subsequently, 30 cc of 0.25% bupivacaine are administered in the depth of the erector spinae, which will remain elevated.

Pectoral Nerve Block type II (PECS II block):

The patient is positioned supine, with the ipsilateral upper limb extended. The clavicular external third line is drawn. In parallel, the lower costal line and the infraclavicular space are highlighted. The probe obtains an image that allows the identification of the pectoralis major and pectoralis minor.

If colour Doppler is added, the acromiothoracic artery is identified and must be avoided.

The needle enters at an angle of 45º from medial to lateral, and 20 cc of 0.25% bupivacaine are administered. Next, needle advances in the interfascial space between the pectoral minor and serratus anterior and 10 cc of 0.25% bupivacaine are administered.

Serratus-Intercostal Fascial Plane Block (SIFP block):

The patient is positioned supine, with the ipsilateral upper extremity at a 90º angle. The fourth, fifth, and sixth intercostal spaces are identified in the mid-axillary line. In coronal section, it is possible to appreciate the subcutaneous cellular tissue, the serratus anterior, and the intercostal muscles.

The needle is introduced at an angle of 30º. From caudal to cranial and resting the needle on the fourth rib, 30 ml of 0.25% bupivacaine are administered between the serratus anterior and lateral intercostal muscles.

Operating room

Next, the patient entered the operating room, and the standard anaesthetic procedure was performed-monitoring with a six-lead electrocardiogram, non-invasive blood pressure, pulse oximetry, and bispectral index. General anaesthesia was induced with intravenous fentanyl 2 mcg/kg, propofol 2-3 mg/kg, and a laryngeal mask adjusted to each patient.

Anaesthetic maintenance was either balanced general anaesthesia with sevoflurane, or total intravenous anaesthesia with propofol in continuous infusion. Ventilation was controlled to maintain normocapnia.

Conventional intravenous analgesia was administered, per protocol was paracetamol 1 g and dexketoprofen 50 mg (in case of allergy to any of these drugs, metamizole 2 g would be administered instead). In addition, as prophylaxis for postoperative nausea and vomiting, ondansetron 4 mg was administered at the end of the intervention.

The anaesthesiologist responsible for the intraoperative period collected data on intraoperative hemodynamic stability, and on the drugs administered.

Postoperative

After anaesthetic delivery, the patients were transferred to the Post-Anaesthesia Recovery (PAR). In the immediate postoperative period, the PAR anaesthesiologist responsible collected the VAS reported by the patient. The postoperative analgesia regimen in PAR consisted of metamizole 2 g, and the responsible physician could prescribe an opioid dose if VAS > 3 at any time during their stay.

After discharge from PAR, if the patient were under the Major Ambulatory Surgery program, the participants would be prescribed postoperative analgesia for 48 hours with paracetamol 1 g every 8 hours and metamizole 575 mg every 8 hours alternately.

In case of hospitalisation, the analgesia regimen consisted of paracetamol 1 g every 8 hours associated with metamizole 2 g every 6 hours. If the patient reported VAS> 3, opioids could be administered according to the individualised care.

Data were collected for the VAS at 24 hours, and the rescue opioids (drug and dose) administered in the first 24 hours. In addition, the length of hospital stay was also collected.

3 months after surgery, the corresponding investigator will collect the VAS score from the patient through a telephonic interview.

1 year after surgery, the corresponding investigator will collect the VAS score, the analgesic treatment needed and location of chronic postoperative pain, from the patient through a telephonic interview. The researcher will collect the analgesic treatment through patient's medical history, and the possible assistance or not by a specialized Pain Unit.

ELIGIBILITY:
Inclusion Criteria:

* Female patient undergoing elective surgery for breast tumour pathology.

Exclusion Criteria:

* Previous breast tumour pathology surgery.
* Breast prosthesis carrier.
* Coagulopathy.
* Pregnancy or lactation.
* Puncture site infection.
* Chest wall deformity.
* Hemodynamically unstable patient.
* Refusal of the patient to undergo locoregional technique.
* The patient refuses to take part in the study or revocation of the Informed Consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Which technique presents less pain in visual analogue scale (VAS score) in the immediate postoperative | Immediate postoperative
  Compare pain management in immediate postoperative period: Which technique presents less pain in visual analogue scale (VAS score), and also comparing this VAS score obtained with the preoperative VAS collected (baseline VAS). VAS is a one-dimensional pain scale (0-no pain; 1-3 mild pain; 4-7 moderate pain; 8-10 severe pain).
Which technique presents less pain in visual analogue scale (VAS score) 24 hours after surgery | 24 hours after surgery
  Compare pain management in postoperative period (24 hours after surgery): Which technique presents less pain in visual analogue scale (VAS score), and also comparing this VAS score obtained with the preoperative VAS collected (baseline VAS). VAS is a one-dimensional pain scale (0-no pain; 1-3 mild pain; 4-7 moderate pain; 8-10 severe pain).
Which technique presents less pain in visual analogue scale (VAS score) 3 months after surgery. | 3 months after surgery
  Compare pain management in postoperative period (3 months after surgery): Which technique presents less pain in visual analogue scale (VAS score), and also comparing this VAS score obtained with the preoperative VAS collected (baseline VAS). VAS is a one-dimensional pain scale (0-no pain; 1-3 mild pain; 4-7 moderate pain; 8-10 severe pain).
Which technique presents less pain in visual analogue scale (VAS score) 1 year after surgery. | 1 year after surgery
  Compare pain management in postoperative period (1 year after surgery): Which technique presents less pain in visual analogue scale (VAS score), and also comparing this VAS score obtained with the preoperative VAS collected (baseline VAS). VAS is a one-dimensional pain scale (0-no pain; 1-3 mild pain; 4-7 moderate pain; 8-10 severe pain).
Rate of participants that required opioid consumption. | 24 hours after surgery
  Which technique requires less opioid use; quantify opioid consumption in milligrams morphine equivalent (MME) and compare opioid consumption between the three study groups.
  Researchers record the opioid use required by patients and the results are converted into MME to make comparison possible.
Rate of participants that required consumption of analgesia 1 year after surgery. | 1 year after surgery
  Comparing the incidence of need of analgesic treatment 1 year after surgery between the three study groups: according to the World Health Organization (WHO) analgesic ladder that patients received one year after surgery.
  WHO analgesic ladder: Step I, treatment with paracetamol and NSAIDs. At step II, treatment with weak opioids; Step III, treatment with a strong opioid; Step IV, interventional pain techniques.

SECONDARY OUTCOMES:
Rate of participants that presented intraoperative hemodynamic alterations | Intraoperative period; an average up to 12 hours.
  Hemodynamics defined by heart rate and non-invasive blood pressure changes that need to be controlled by drugs.
  YES: patients present hemodynamic alterations (Mean arterial pressure <65 mmHg or >20% variation; heart rate >100 heart beats per minute).
  NO: patients do not present any hemodynamic alterations.
The Length (number of hours) of Hospital Stay: comparison between the three study groups. | Number of hours from hospitalization; from Major Outpatient Surgery (0 hours) to 7 days (168 hours) Hospital Stay
  Quantify in hours the hospital stay length and compare results between the three study groups.
Assistance by Pain Unit: comparison between the three study groups. | 1 year after surgery
  Analyze how many patients with chronic postsurgical pain are being followed by the Pain Unit.Compare the assistance needed between the three study groups
Compare the incidence of location of chronic postoperative pain between the three study groups. | 1 year after surgery
  Breast CPP: patients with pain in the breast area and chest wall. Shoulder CPP: patients with ipsilateral shoulder and/or upper limb pain. Breast & Shoulder CPP: patients who unify both locations described. Comparing locations incidence in three groups of study.

CONTACTS AND LOCATIONS:
Overall Officials: Jose De Andrés Ibáñez, MD, PhD, Principal Investigator — jose.andres@uv.es
Locations (1):
- José De Andrés Ibáñez, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No